CLINICAL TRIAL: NCT00164658
Title: Evaluating Tools for Health Promotion and Disease Prevention
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Case Western Reserve University (Other); American Academy of Family Physicians National Research Network (Network); Evanston Northwestern Healthcare Research Institute (Unknown); University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CDC-OGDP-4444; U36/CCU319276-MM-0630; U50/CCU300860-TS-1216; U36/CCU319276-MM-0789
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2010-01

CONDITIONS: Coronary Heart Disease; Stroke; Diabetes; Breast Cancer; Ovarian Cancer; Colorectal Cancer
Keywords: family history; familial risk; behavior change
MeSH Terms: conditions — Coronary Disease; Stroke; Diabetes Mellitus; Breast Neoplasms; Ovarian Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Familial risk assessment and personalized prevention messages

SUMMARY:
The study will evaluate the effect of familial risk assessment and prevention prompts tailored to familial risk on health behaviors and use of preventive services among adults who are members of primary care practices in the U.S.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the clinical utility of a new family history tool, Family Healthware™ by determining whether family history risk assessment and personalized prevention messages have any impact on health behaviors and use of medical services. The hypothesis to be tested is that patients who are provided with personalized prevention messages based on an assessment of their family history of disease will be more motivated to make behavior changes and use preventive health services than patients who do not have their family history assessed and who receive only generalized (not personalized) prevention messages. An additional hypothesis, tested when participants see their primary care physician during the study, is that providing a copy of the graphical family history, risk and prevention messages to the patient's physician will increase delivery of recommended preventive services (screening, referral, and health habit advice).

The study will consist of enrolling approximately 8360 patients aged 35-65 years who attend primary care practices that are part of research networks affiliated with the three research centers. The practices will be randomized into two groups. Patients in practices randomized to Group 1 will complete a pre-test and the family history tool, and will receive personalized prevention messages based on their level of familial risk and current risk behaviors. After six months, Group 1 patients will complete a post-test. Patients in Group 2 will complete the pre-test and receive standard prevention messages (appropriate for sex) about maintaining good health and preventing disease. After 6 months Group 2 patients will complete the post-test and the family history tool. The pre- and post-test will include assessment of risk factors, use of medical services (especially preventive services), interest in modifying health behaviors, risk perceptions, etc. The analysis will compare changes in health behaviors between patients in Groups 1 and 2 and will also examine differences by familial risk strata (average, moderate, high).

ELIGIBILITY:
Inclusion Criteria:

* member of participating primary care practice network
* able to provide informed consent
* able to complete data assessment tools in English

Exclusion Criteria:

* diagnosis of CHD, stroke, diabetes, breast cancer, ovarian cancer, or colorectal cancer
* currently pregnant
* evidence of cognitive impairment

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8400 (Estimated)
Dates: Start 2005-09; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Change in stage of adoption of health behaviors and referral for additional screening and follow up for high risk participants at 6 month post evaluation

SECONDARY OUTCOMES:
Primary care physicians' provision of preventive services in response to family medical history.

CONTACTS AND LOCATIONS:
Overall Officials: Louise S Acheson, MD, MS, Principal Investigator — Case Western Reserve University Department of Family Medicine & CWRU/UHC Comprehensive Cancer Center; Wendy S Rubinstein, MD, PhD, Principal Investigator — Evanston Northwestern Healthcare Research Institute; Suzanne M O'Neill, MA, MS, PhD, Principal Investigator — Evanston Northwestern Healthcare Research Institute; Mack T Ruffin IV, MD, MPH, Principal Investigator — University of Michigan
Locations (3):
- United States (3):
  - Evanston Northwestern Healthcare (ENH) internal medicine, family practice, and OB/GYN practices, Evanston, Illinois
  - American Academy of Family Physicians National Research Network (AAFP-NRN)., Leawood, Kansas
  - Great Lakes Research into Practice Network (GRIN), Ann Arbor, Michigan

REFERENCES:
- [Derived] Wang C, Sen A, Plegue M, Ruffin MT 4th, O'Neill SM, Rubinstein WS, Acheson LS; Family Healthware Impact Trial (FHITr) Group; Family Healthware Impact Trial FHITr Group. Impact of family history assessment on communication with family members and health care providers: A report from the Family Healthware Impact Trial (FHITr). Prev Med. 2015 Aug;77:28-34. doi: 10.1016/j.ypmed.2015.04.007. Epub 2015 Apr 19. PMID 25901453
- [Derived] Wang C, Sen A, Ruffin MT 4th, Nease DE Jr, Gramling R, Acheson LS, O'Neill SM, Rubinstein WS; Family Healthware Impact Trial (FHITr) Group. Family history assessment: impact on disease risk perceptions. Am J Prev Med. 2012 Oct;43(4):392-8. doi: 10.1016/j.amepre.2012.06.013. PMID 22992357
- [Derived] Dorman JS, Valdez R, Liu T, Wang C, Rubinstein WS, O'Neill SM, Acheson LS, Ruffin MT 4th, Khoury MJ. Health beliefs among individuals at increased familial risk for type 2 diabetes: implications for prevention. Diabetes Res Clin Pract. 2012 May;96(2):156-62. doi: 10.1016/j.diabres.2011.12.017. Epub 2012 Jan 17. PMID 22257420
- [Derived] Ruffin MT 4th, Nease DE Jr. Using patient monetary incentives and electronically derived patient lists to recruit patients to a clinical trial. J Am Board Fam Med. 2011 Sep-Oct;24(5):569-75. doi: 10.3122/jabfm.2011.05.100169. PMID 21900440
- [Derived] O'Neill SM, Rubinstein WS, Wang C, Yoon PW, Acheson LS, Rothrock N, Starzyk EJ, Beaumont JL, Galliher JM, Ruffin MT 4th; Family Healthware Impact Trial group. Familial risk for common diseases in primary care: the Family Healthware Impact Trial. Am J Prev Med. 2009 Jun;36(6):506-14. doi: 10.1016/j.amepre.2009.03.002. PMID 19460658